CLINICAL TRIAL: NCT05371509
Title: Novel Myofunctional Water Bottle to Reduce OSA and Snoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Remastered Sleep LLC (Unknown)
Responsible Party: Principal Investigator, Umesh Goswami, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-001883; R43HL160368 (NIH)
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea; Snoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring | interventions — Myofunctional Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Myofunctional therapy (MT) nozzle (Experimental): Subjects diagnosed with mild to moderate obstructive sleep apnea will receive a water bottle with a myofunctional therapy (MT) nozzle to use daily
  Interventions: Device: Myofunctional therapy (MT) nozzle
- Placebo nozzle (Placebo Comparator): Subjects diagnosed with mild to moderate obstructive sleep apnea will receive a water bottle with a placebo nozzle to use daily
  Interventions: Other: Placebo nozzle

INTERVENTIONS:
Device: Myofunctional therapy (MT) nozzle — Water bottle nozzle designed to allow the user to repeatedly perform the tongue suction, tongue press, and swallow exercise movements while also providing targeted resistance to train and improve tongue, soft palate, and pharyngeal muscle strength and endurance.
  Arms: Myofunctional therapy (MT) nozzle
Other: Placebo nozzle — The placebo bottle nozzle will look similar to the MT nozzle; but is not expected to function the same as the MT nozzle.
  Arms: Placebo nozzle

SUMMARY:
This research study is being done to determine whether the repetition and resistance from the daily use of the myofunctional therapy (MT) nozzle will improve obstructive sleep apnea and primary snoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate obstructive sleep apnea with Apnea Hypopnea Index 5-29 events/hour confirmed within last 2 years with an in-lab diagnostic polysomnography or home sleep apnea test.
* Ownership of a smartphone and willingness to use a smartphone application to automatic log daily water intake.
* Willingness and ability to discontinue the currently prescribed OSA treatment for at least 3 days prior to testing.
* Age greater than or equal to 18 years.
* Participants willing to travel to the Rochester area for the Speech and Language Pathologist exam

Exclusion Criteria:

* Significant weight change (10% change in body weight in Kg) from the time of the OSA diagnosis until the study initiation.
* Persistent excessive daytime sleepiness (Epworth Sleepiness scale > 10), despite treatment of OSA
* Significant medical comorbidities requiring restricted oral fluid intake - decompensated heart failure, end stage renal disease, end stage liver disease, hyponatremia (S. Na <130 mg/dl), nocturia > times/night.
* Significant mental health comorbidities including history of psychogenic polydipsia, obsessive-compulsive behavior, current suicidal ideation and uncontrolled anxiety.
* Unable or unwilling to participate in study procedures.
* Previous upper airway surgeries significantly modifying upper airway anatomy.
* Known congenital or acquired diseases significantly affecting upper airway anatomy.
* BMI >40 kg/m^2.
* Currently treating OSA with hypoglossal nerve stimulator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Umesh Goswami, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 subjects were enrolled in the study and 1 subject withdrew prior to randomization.
Groups:
- Myofunctional therapy (MT) nozzle: Subjects diagnosed with mild to moderate obstructive sleep apnea received a water bottle with a myofunctional therapy (MT) nozzle to use daily
  Myofunctional therapy (MT) nozzle: Water bottle nozzle designed to allow the user to repeatedly perform the tongue suction, tongue press, and swallow exercise movements while also providing targeted resistance to train and improve tongue, soft palate, and pharyngeal muscle strength and endurance.
- Placebo nozzle: Subjects diagnosed with mild to moderate obstructive sleep apnea receivede a water bottle with a placebo nozzle to use daily
  Placebo nozzle: The placebo bottle nozzle looked similar to the MT nozzle; but is not expected to function the same as the MT nozzle.
Period: Overall Study
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myofunctional Therapy (MT) Nozzle | Placebo Nozzle | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.9) | 51.38 (10.23) | 55.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 8 | 15 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Therapy
Description: The was measured as the number of days subjects met their daily water consumption goal. Subjects were asked to hit their daily water consumption goal 5 days per week for 8 weeks.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
Number analyzed (Participants) | 20 | 21
days | 18.4 (16.4) | 26.1 (15.2)

2. Primary Outcome: Change in Quality of Life
Description: Measured using the Calgary Sleep Apnea Quality of Life Index (SAQLI) questionnaire which assesses the quality of life in individuals with obstructive sleep apnea. It has a score between 1 and 7 on five different domains with total scores ranging from 7 to 42, with higher scores indicating a worse quality of life.
Time Frame: Baseline, Day 60
Population: Five subjects in the myofunctional therapy arm and 7 subjects in the placebo arm did not complete the SAQLI at both baseline and day 60, therefore the change in quality of life was unable to be reported for those subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
Number analyzed (Participants) | 15 | 14
score on a scale | -0.02 (1.74) | 0.34 (0.78)

3. Secondary Outcome: Change in Apnea Hypopnea Index (AHI)
Description: The Apnea Hypopnea Index (AHI) assesses the severity of sleep apnea by measuring the number of apneas (complete cessation of breathing for at least 10 seconds) and hypopneas (partial reductions in airflow) that occur during an hour of sleep. For this study AHI was measured through use of the WatchPAT One device.
Time Frame: Baseline, Day 60
Population: There was an error in the WatchPAT device data in 2 subjects in the Myofunction therapy arm and 5 in the placebo arm causing there to be no data for change in AHI for those subjects.
Measure: Mean (Standard Deviation); unit: AHI
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
Number analyzed (Participants) | 18 | 16
AHI | -0.9 (6.3) | 2.7 (6.8)

4. Secondary Outcome: Change in Myofunction Assessment
Description: Myofunction assessment was done using the Iowa Oral Performance Instrument (IOPI) which involves measuring the strength and endurance of the tongue which aids in the diagnosis and treatment of obstructive sleep apnea. The assessment is done on both the anterior (front) and posterior (back) side of the tongue and measured in kilopascals (kPa). Normal values range from 40-80 kPa, with higher values indicating higher tongue strength and endurance.
Time Frame: Baseline, Day 60
Population: 2 subjects in the placebo arm did not complete the myofunction assessment at both the baseline and day 60 visit therefore no data was available to calculate change in the myofunctional assessment for those subjects.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
Number analyzed (Participants) | 20 | 19
kPa
  IOPI Anterior | 0.6 (6.2) | -1.3 (7.2)
  IOPI Posterior | 1.3 (7.3) | 0.7 (7.0)

5. Secondary Outcome: Change in Oxygen Saturation (SpO2)
Description: SpO2 was measured using the WatchPat One device. SpO2 is a measurement of the percentage of oxygen-bound hemoglobin in the blood.
Time Frame: Baseline; 60 Days
Population: There was an error in the WatchPAT device data in 1 subject in the Myofunction therapy arm and 5 in the placebo arm causing there to be no data for change in SpO2 for those subjects.
Measure: Mean (Standard Deviation); unit: percent of oxygen in blood
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
Number analyzed (Participants) | 19 | 16
percent of oxygen in blood | 0.37 (0.84) | -0.07 (1.00)

6. Secondary Outcome: Change in Snoring Intensity
Description: Snoring intensity was measured through a questionnaire that was administered to the subject's bed partner that asked "Over the past few days, how would you describe your spouse/bed partner's snoring?" Scores ranged from -3 (worst) to +3 (best) with higher scores indicating lower snoring intensity.
Time Frame: Baseline; Day 60
Population: 4 subjects in the Myofunctional Therapy arm and 13 subjects in the placebo arm did not complete the snoring intensity question at both the baseline and day 60 visit therefore no data was available to calculate change in the snoring intensity for those subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
Number analyzed (Participants) | 16 | 8
score on a scale | 0.38 (0.81) | 0.25 (1.04)

7. Secondary Outcome: Change in Snoring Frequency
Description: Snoring Frequency was measured through a questionnaire that was administered to the subject's bed partner that asked "Over the past few days, how often did you notice your bed partner's snoring?" Scores ranged from -4 (worst) to +4 (best) with higher scores indicating lower snoring frequency.
Time Frame: Baseline; Day 60
Population: 3 subjects in the Myofunctional Therapy arm and 12 subjects in the placebo arm did not complete the snoring frequency question at both the baseline and day 60 visit therefore no data was available to calculate change in the snoring frequency for those subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
Number analyzed (Participants) | 17 | 9
score on a scale | 0.65 (1.00) | 0.89 (1.90)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 3 months.
Arm/Group | Myofunctional therapy (MT) nozzle | Placebo nozzle
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT05371509/Prot_001.pdf
  • Informed Consent Form (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT05371509/ICF_000.pdf